CLINICAL TRIAL: NCT02835651
Title: Effects of C16:0 Versus C18:0 on HDL Metabolism and Other Cardiometabolic Risk Markers: A Dietary Intervention Study in Healthy Normal-weight and Overweight Subjects
Brief Title: Saturated Fatty Acids and HDL Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 15-3-052
Record Dates: First submitted 2016-05-18; First posted 2016-07-18 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-03

CONDITIONS: Dyslipidemia
Keywords: Palmitic acid; Stearic acid; HDL-metabolism; Human intervention study
MeSH Terms: conditions — Dyslipidemias | interventions — Palmitic Acid; stearic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Palmitic acid (Experimental): Diet rich in palmitic acid
  Interventions: Dietary Supplement: Palmitic acid
- Stearic acid (Experimental): Diet rich in stearic acid
  Interventions: Dietary Supplement: Stearic acid

INTERVENTIONS:
Dietary Supplement: Palmitic acid — Experimental products are enriched with C16:0
  Arms: Palmitic acid
Dietary Supplement: Stearic acid — Experimental products are enriched with C18:0
  Arms: Stearic acid

SUMMARY:
The purpose of this study is to determine whether palmitic acid (C16:0) and stearic acid (C18:0) have different effects on HDL metabolism during the fasted state.

DETAILED DESCRIPTION:
Study design:

Double blind, randomized, cross-over study with two different diets: one diet will be high in palmitic acid (C16:0) and the other diet will be high in stearic acid (C18:0). Subjects will receive both diets for 4 weeks with a wash-out period of 4-6 weeks in between. Contrast in the intakes of palmitic acid and stearic acid is 6% of energy. A postprandial test will be carried out at the end of each dietary period.

Study population:

Accounting for a dropout rate of 20%, 40 healthy men and postmenopausal women, aged between 45 and 70 year, having a BMI (body mass index) between ≥ 18.0 and ≤ 30.0 kg/m2 will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and post-menopausal women (post-menopausal for at least one year) as judged by study physician
* BMI ≥ 18.0 and ≤ 30.0 kg/m2
* Aged between 45 and 70 years
* Willing to comply to study protocol during study
* Having a general practitioner
* Agreeing to be informed about medically relevant personal test-results by a physician
* Informed consent signed
* Accessible veins on arms as determined by examination at screening

Exclusion Criteria:

* Having a medical condition which might impact study measurements
* Use of over-the-counter and prescribed medication, which may interfere with study measurements
* Use of oral antibiotics in 40 days or less prior to the start of the study;
* Use of food supplements or plant-sterol/stanol-enriched foods or supplements in the three months prior to the screening and/or during the study;
* Reported alcohol consumption ≥ 10 units/week (female) or ≥ 14 units/week (male);
* Reported intense sporting activities ≥ 10 hours/week;
* Reported weight loss or gain of 3 kg or more during a period of 2 months prior to screening
* Regular smokers (at least one cigarette (or equivalent) daily or >7 cigarettes (or equivalent) weekly. Smokers who cannot comfortably restrain from smoking for up to 2 days will also be excluded
* Reported dietary habits: medically prescribed diet, allergy/intolerance to test products that will be provided during the study
* Blood donation in the past 3 months
* Drug abuse
* Reported participation in another nutritional or biomedical trial 3 months prior to screening
* Fasting triacylglycerol concentrations at screening: ≥ 4.5 mmol/L
* Serum lipids: treatment recommended according to the "Multidisciplinary guidelines Cardiovascular risk management"
* Fasting HbA1c ≥ 48 mmol/mol (or 6.5%)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Cholesterol efflux capacity after dietary period high in palmitic acid compared to dietary period high in stearic acid | Cholesterol efflux is measured during fasted state at day 0, day 25 and day 28 of each intervention period.
  J774 Macrophages will be used to measure ex vivo cholesterol efflux capacity of HDL particles after a diet enriched with C16:0 or C18:0. Change in ex vivo cholesterol efflux capacity between the diets will be assessed using a linear mixed model with subject as random factor and day 0 as co-variant.

SECONDARY OUTCOMES:
Change in fasted lipid metabolism markers between dietary period high in palmitic acid and dietary period high in stearic acid | Markers for lipid metabolism will be measured during fasted state at day 0, day 14, day 25 and day 28 of each intervention period
  Markers include fasting LDL-C [mmol/L], HDL-C [mmol/L], total cholesterol [mmol/L], non-HDL cholesterol [mmol/L] and triacylglycerol [mmol/L] concentrations. Change between diets will be assessed using a linear mixed model with subject as random factor and day 0 as co-variant.
Change in fasted lipid ratios between dietary period high in palmitic acid and dietary period high in stearic acid | Markers for lipid metabolism will be measured during fasted state at day 0, day 14, day 25 and day 28 of each intervention period
  Markers include fasting total cholesterol to HDL-C ratio and LDL-C to HDL-C ratio. Change between diets will be assessed using a linear mixed model with subject as random factor and day 0 as co-variant.
Change in fasted apolipoproteins between dietary period high in palmitic acid and dietary period high in stearic acid | Apolipoproteins will be measured during fasted state at day 0, day 14, day 25 and day 28 of each intervention period
  Apolipoproteins include fasting ApoA1 [μg/mL] and ApoB100 [μg/mL]. Change between diets will be assessed using a linear mixed model with subject as random factor and day 0 as co-variant.
Change in postprandial triacylglycerol levels between dietary period high in palmitic acid and dietary period high in stearic acid | Triacylglycerol [mmol/L] is measured during postprandial state at day 28 (0 to 480 minutes after meal intake) of each intervention period
  Change between diets will be assessed using a linear mixed model with subject as random factor and day 0 as co-variant.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van Rooijen MA, Plat J, Zock PL, Blom WAM, Mensink RP. Effects of two consecutive mixed meals high in palmitic acid or stearic acid on 8-h postprandial lipemia and glycemia in healthy-weight and overweight men and postmenopausal women: a randomized controlled trial. Eur J Nutr. 2021 Oct;60(7):3659-3667. doi: 10.1007/s00394-021-02530-2. Epub 2021 Mar 17. PMID 33733339
- [Derived] van Rooijen MA, Plat J, Blom WAM, Zock PL, Mensink RP. Dietary stearic acid and palmitic acid do not differently affect ABCA1-mediated cholesterol efflux capacity in healthy men and postmenopausal women: A randomized controlled trial. Clin Nutr. 2021 Mar;40(3):804-811. doi: 10.1016/j.clnu.2020.08.016. Epub 2020 Aug 27. PMID 32900520